CLINICAL TRIAL: NCT04687761
Title: A Phase I-II, Multicentre, Open Label Clinical Trial to Assess the Safety and Tolerability of the Combination of Low-dose Cytarabine or Azacitidine, Plus Venetoclax and Quizartinib in Newly Diagnosed Acute Myeloid Leukemia Patients Aged Equal or More Than 60 Years Old Ineligible for Standard Induction Chemotherapy
Brief Title: Clinical Trial to Assess the Safety and Tolerability of the Combination of Low-dose Cytarabine or Azacitidine Plus Venetoclax and Quizartinib in Newly Diagnosed AML Patients Aged Equal or More Than 60 Years Old
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VEN-A-QUI
Record Dates: First submitted 2020-11-17; First posted 2020-12-29 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Leukemia, Myeloid, Acute; De Novo; Age More 60yr
Keywords: Acute myeloid Leukaemia; Newly Diagnosed
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax; quizartinib; Cytarabine

STUDY DESIGN:
Intervention Model Description: Phase 1: Study treatment will start at level 1 and therapeutic level will be escalated or descalated depending on the apparition of DLT. DLT will be monitored during cycle 1 and it is defined as any grade 3-4 related extrahematological toxicity or grade 4 neutropenia not recovered on day 56 since C1D1 not attributable to persistent leukemia.
  Phase I will consist of two parallel dose escalation cohorts, with consecutive assignment to each group (first patient will be assigned to AZA-based schedule, second to LDAC-based, third to AZA-based, etc).
  Phase II includes two treatment arm groups (AZA-based RP2D vs. LDAC-based RP2D). Patients will be enrolled at diagnosis, within a maximum 28 days screening period, will be assessed for eligibility and therefore randomized to follow the assigned treatment arm (open label design). All screening activities will be performed after patient's informed consent form is signed. Patients will start the assigned regimen 48h maximum after randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZA-Based (Experimental): Azacitidine 75 mg/m2/daily SC on a 5-on/2-off [weekend]/2-on schedule in 28-day cycle plus Venetoclax (ramp-up) 400 mg/daily oral, days 1 to 28 plus Quizartinib phase I/RP2D mg/daily oral, days 8 to 14-28.
  If 1 DLT is observed among these 3 patients, additional 3 subjects will receive the level 2 dose, and it will be recommended in the absence of DLT between them. If >1 DLT occurs in these 6 level 2 patients, the dose administered in the level 1 will be the RP2D of the AZA-based schedule.
  AZA and Venetoclax doses will remain the same in all levels and only the dose of Quizartinib will be modificated according to the following table:
  Escalation-Quizartinib dose-Quizartinib duration; Level-2 -30 mg/daily-Days 8 to 14; Level-1 -30 mg/daily-Days 8 to 21; Level1-40 mg/daily Days 8 to 28; Level2-60 mg/daily-Days 8 to 28.
  In phase II, patients randomized to this arm, will receive the recommended phase 2 dose (RP2D) regimen of AZA + Venetoclax + Quizartinib regimen (30 patients).
  Interventions: Drug: Azacitidine; Drug: Venetoclax; Drug: Quizartinib
- LDAC-Based (Experimental): Low-dose subcutaneous cytarabine 20 mg/m2/daily SC, days 1 to 10 plus Venetoclax (ramp-up) 600 mg/daily oral, days 1 to 28 plus Quizartinib phase I/RP2D mg/daily oral, days 8 to 14-28.
  If 1 DLT is observed among these 3 patients, additional 3 subjects will receive the level 2 dose, and it will be recommended in the absence of DLT between them. If >1 DLT occurs in these 6 level 2 patients, the dose administered in the level 1 will be the RP2D of the LDAC-based schedule.
  LDAC and Venetoclax doses will remain the same in all levels and only the dose of Quizartinib will be modificated according to the following table:
  Escalation-Quizartinib dose-Quizartinib duration; Level-2 -30 mg/daily-Days 8 to 14; Level-1 -30 mg/daily-Days 8 to 21; Level1-40 mg/daily-Days 8 to 28; Level2-60 mg/daily-Days 8 to 28.
  In phase II, patients randomized to this arm, will receive the recommended phase 2 dose (RP2D) regimen of LDAC + Venetoclax + Quizartinib regimen (30 patients).
  Interventions: Drug: Cytarabine; Drug: Venetoclax; Drug: Quizartinib

INTERVENTIONS:
Drug: Azacitidine — AZA 75 mg/m2/daily SC days 1 to 7 or on a 5-on/2-off [weekend]/2-on schedule in 28-day cycle
  Arms: AZA-Based
Drug: Venetoclax — Venetoclax (ramp-up) 400 mg/daily oral days 1 to 28
  Arms: AZA-Based
Drug: Quizartinib — Quizartinib 40 mg/daily oral, days, 8 to 28
  Arms: AZA-Based
Drug: Cytarabine — Low-dose subcutaneous cytarabine (LDAC) 20 mg/m2/daily SC, days 1 to 10
  Arms: LDAC-Based
Drug: Venetoclax — Venetoclax (ramp-up) 600 mg/daily oral, days 1 to 28
  Arms: LDAC-Based
Drug: Quizartinib — Quizartinib 40 mg/daily oral, days 8 to 28
  Arms: LDAC-Based

SUMMARY:
A phase I-II trial based on the combination of three drugs regimen LDAC or Azacitidine + Venetoclax + Quizartinib that in this population could be well tolerated by a sequential type administration. The first objective is to achieve rapid control of the disease, using two different schemes, one based in Azacitidine and the other in LDAC, by dose escalation in phase I of the trial. The second goal is to prevent relapse through a maintenance schedule. Phase II will study the efficacy and safety of the recommended dose for Phase II

DETAILED DESCRIPTION:
The prognosis of AML in elderly patients remain very poor and without significant advances in last decades. AML is a heterogeneous disease in which many altered molecular pathways could contribute to the disease. Thus, curative approaches have been based on highly eradicating regimens using high-dose chemotherapy. However, the low rate of CRs and the high rate of deaths due to toxicity and relapses in elderly patients should stimulate the development of new regimens that overcome these therapeutic obstacles. In recent years, there are a series of new drugs under development that allow the design of sequential combination therapies in this vulnerable population. These drugs have an acceptable toxicity profile and are apparently effective in monotherapy or even in combination, being able to improve the CR rate in this population. The investigators hypothesize that the combination of two targeted drugs that have different mechanisms of action could be capable of breaking the viability of leukemic cells as well as their proliferative qualities, and therefore prolong survival. In this way, the combined action of a pro-apoptotic agent (Venetoclax) and an antiproliferative agent (Quizartinib) could produce a powerful antileukemic effect, preventing the adaptive escape mechanisms of leukemic cells. The investigators have designed a phase I-II trial based on the combination of three drugs regimen LDAC or Azacitidine + Venetoclax + Quizartinib that in this population could be well tolerated by a sequential type administration. The first objective is to achieve rapid control of the disease, using two different schemes, one based in Azacitidine and the other in LDAC, by dose escalation in phase I of the trial. The second goal is to prevent relapse through a maintenance schedule. Phase II will study the efficacy and safety of the recommended dose for Phase II.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed AML.
2. Morphological diagnosis of AML (WHO criteria 2008).
3. Patient must be considered be ineligible for treatment with a standard cytarabine and anthracycline induction regimen due to age or co-morbidities defined by the following criteria: 3.1. ≥ 71 years of age; 3.2. ≥ 60 to 70 years of age with at least one of the following co-morbidities:

   * ECOG Performance Status of 2 or 3;
   * Cardiac history of CHF requiring treatment or Ejection Fraction ≤ 55% or chronic stable angina;
   * DLCO ≤ 65% or FEV1 ≤ 65% or significant history of chronic pulmonary obstructive;
   * Creatinine clearance ≥ 30 mL/min to < 50 ml/min
   * Moderate hepatic impairment with total bilirubin, SGPT or SGOT > 1.5 to ≤ 3.0 × ULN
   * Non active/controlled prior neoplastic disease
   * Any other patient´s comorbidity or disease condition that the physician judges to be incompatible with intensive chemotherapy must be reviewed and approved by the Trial Coordinators before study enrollment (e.g, prior MDS or MPS, high-risk cytogenetics)
4. ECOG performance status ≤ 3.
5. Male subjects who are sexually active, must agree, from Study Day 1 through at least 120 days after the last dose of study drug, to practice the protocol specified contraception (see Section 0).
6. Female subjects must be either postmenopausal for at least 1 year before screening OR permanently surgical sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy) OR Women of Childbearing Potential (WOCBP) must agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug (female and male condoms should not be used together), or Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception). Female subjects of childbearing potential must have negative results for pregnancy test performed and must not be lactating and breastfeeding.
7. Subject must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC) prior to the initiation of any screening or study specific procedures, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

1. Age <60 years.
2. Genetic diagnosis of acute promyelocytic leukemia.
3. Treated (excluding surgery or hormone-therapy) for another malignancy within 6 months before randomization or previously diagnosed with another malignancy and have any evidence of disease which may compromise the administration of investigational treatment schedule.
4. Presence of any severe psychiatric disease or physical condition that, according to the physician´s criteria, contraindicates the inclusion of the patient into the clinical trial.
5. Serum creatinine ≥ 2.5 mg/dL or creatinine clearance < 30 mL/min (unless it is attributable to AML activity).
6. Bilirubin, SGPT or SGOT > 3 times the upper normal limit (unless it is attributable to AML activity).
7. WBC> 50 x 109/L. Subject should have white blood cell count <50 × 109/L before starting therapy. Patients who are cytoreduced with leukapheresis or with hydroxyurea may be enrolled if they meet the eligibility criteria before starting therapy.
8. Contraindications for Quizartinib or Venetoclax.
9. History of known CNS leukemia, including cerebrospinal fluid positive for AML blasts.
10. Prior treatment with any investigational drug or device within 30 days prior to Randomization (within 2 weeks for investigational or approved immunotherapy) or currently participating in other investigational procedures
11. Prior treatment with other FLT3-ITD or BCL-2 inhibitors.
12. Known uncontrolled or significant cardiovascular disease, including any of the following:

    1. Bradycardia of less than 50 beats per minute, unless the subject has a pacemaker;
    2. QTcF interval >450 msec;
    3. Diagnosis of or suspicion of long QT syndrome (including family history of long QT syndrome);
    4. Systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg;
    5. History of clinically relevant ventricular arrhythmias (eg, ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes);
    6. History of second (Mobitz II) or third degree heart block (subjects with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker);
    7. History of uncontrolled angina pectoris or myocardial infarction within 6 months prior to Screening;
    8. History of New York Heart Association Class 3 or 4 heart failure;
    9. Known history of left ventricular ejection fraction (LVEF) ≤45% or less than the institutional lower limit of normal;
    10. Complete left bundle branch block;
13. Prior therapy for AML (except hydroxiurea).
14. Subject enrolling into a dose-escalation cohort must not have received a known strong or moderate inducer or inhibitor of cytochrome P450 (CYP) 3A within 7 days before the first Quizartinib or Venetoclax dose. Subject enrolling into a safety expansion cohort must not have received a known strong or moderate inducer or strong inhibitor of CYP3A within 7 days before the first Quizartinib or Venetoclax dose.
15. Subject must not have consumed grapefruit, grapefruit products, Seville oranges (including marmalade-containing Seville oranges), or star fruit within 3 days before anticipated first dose of Venetoclax and must consent not to consume through the last dose of Venetoclax.
16. Active acute or chronic systemic fungal, bacterial, or viral infection not well controlled by antifungal, antibacterial or antiviral therapy at physician discretion;
17. Known active clinically relevant liver disease (eg, active hepatitis B, or active hepatitis C)
18. Known history of human immunodeficiency virus (HIV).
19. History of hypersensitivity to any excipients in the Quizartinib, Venetoclax or other study medication.
20. Non mutated FLT3-ITD subjects will be considered ineligible during the randomized Phase II after 48 non mutated FLT3-ITD subjects have been randomized.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-11-04 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Phase I: Recommended phase 2 dose (RP2D) | Approximately 6 months after first patient first visit (FPFV)
  Recommended phase 2 dose (RP2D) of AZA based and LDAC based triple combination with Quizartinib and Venetoclax schedules
Phase II: CR/Cri rate of AZA based and LDAC based | Aproximatey 3 years after FPFV
  CR/CRi rate of AZA based and LDAC based triple combination with Quizartinib and Venetoclax schedules.
  Patients will receive 4 consecutive cycles of treatment (approximately every 28 days). After the first 4 cycles, depending on the response and tolerance to treatment, the patient will continue receiving treatment in maintenance cycles until one of these situations occurs: disease progression, lack of clinical benefit, hematological relapse, unacceptable toxicity.

SECONDARY OUTCOMES:
CR/CRi rate | After cycle 1 and after cycle 4, being each cycle of 28 days
  To evaluate the CR/CRi rate after 1 and 4 cycles of AZA based and LDAC based triple combination with Quizartinib and Venetoclax schedules.
Overall survival (OS) | Through study completion: 2 years after the last patient has been enrolled into the study, an average of 48 months.
  Overall survival will be defined as the number of days from the start of treatment to the date of death. Subjects that have not died will be censored at the last known date to be alive. To estimate 1, 2 and 3 years event-free, disease-free, and relapse-free survival, as well as on the cumulative incidence of relapse.
Overall hematologic and non-hematologic toxicity | Through study completion: 2 years after the last patient has been enrolled into the study, an average of 48 months.
  To evaluate the safety and tolerability of AZA based and LDAC based triple combination with Quizartinib and Venetoclax schedules (overall hematologic and non-hematologic toxicity).
Event-free survival (EFS) | 1, 2 and 3 years.
  EFS will be defined as the time from enrollment until the date of progressive disease, relapse from CR or CRi, failure to achieve CR or CRi at 6 months after initiation of treatment, or death from any cause. If a specified event does not occur, subjects will be censored at the date of last disease follow-up. Data for subjects without any disease assessments performed after enrollment will be censored at the date of enrollment.
Disease-free survival (DFS) | 1, 2 and 3 years.
  DFS will be defined as the time from achieving CR or CRi until the date of relapse or death from any cause, whichever occurs first.
Relapse-free survival (RFS) | 1, 2 and 3 years.
  RFS will be defined as the time from achieving CR or CRi until the date of relapse.
Cumulative incidence of relapse | 1, 2 and 3 years.
  Estimation of cumulative incidence of relapse
Impact on the quality of life assessed by EuroQoL Group EQ-5D-5L | At the screening, after cycle 2, after cycle 6, and after cycle 12, being each cycle of 28 days; and through study completion, an average of 48 months.
  The impact on the quality of life will be assessed using the EuroQoL Group EQ-5D-5L instrument.
Impact on the quality of life assessed by EORTC QLQ-C30 | at the screening, after 6 cycles, after 12 cycles since start of therapy, being each cycle of 28 days; and through study completion, an average of 48 months
  The impact on the quality of life will be assessed using the EORTC QLQ-C30 instrument.
Use of medical resources during treatment phase | At the end of treatment phase: after cycle 4, being each cycle of 28 days.
  To evaluate the impact on the use of medical resources during treatment phase (ie, antibiotics, transfusions, duration of hospitalization, need of central venous line, use of strong or moderate CYP3A inhibitors and moderate CYP3A inducers).
Quality of CR | After cycle 1, cycle 4 and then every 3 cycles during the first 2 years after start of the therapy (each cycle of 28 days).
  To evaluate the quality of CR (by study of minimal residual disease percentages in the bone marrow (BM) using multiparametric flow cytometry [MPFC] and NGS-MRD).
CRh rate | Through study completion: 2 years after the last patient has been enrolled into the study, an average of 48 months.
  To evaluate the CRh rate in AZA based and LDAC based triple combination with Quizartinib and Venetoclax schedules.
Early mortality | First 30 and 60 days
  To evaluate early mortality rate in AZA based and LDAC based triple combination with Quizartinib and Venetoclax schedules.
CR/Cri rate of AZA based and LDAC based, in secondary AML subset | Through study completion: 2 years after the last patient has been enrolled into the study, an average of 48 months.
  CR/CRi rate of AZA based and LDAC based triple combination with Quizartinib and Venetoclax schedules.
CR/Cri rate of AZA based and LDAC based, in CBF subset | Through study completion: 2 years after the last patient has been enrolled into the study, an average of 48 months.
  CR/CRi rate of AZA based and LDAC based triple combination with Quizartinib and Venetoclax schedules.
CR/Cri rate of AZA based and LDAC based, in FLT3-ITD subset | Through study completion: 2 years after the last patient has been enrolled into the study, an average of 48 months.
  CR/CRi rate of AZA based and LDAC based triple combination with Quizartinib and Venetoclax schedules.
CR/Cri rate of AZA based and LDAC based, in NPM1 subset | Through study completion: 2 years after the last patient has been enrolled into the study, an average of 48 months.
  CR/CRi rate of AZA based and LDAC based triple combination with Quizartinib and Venetoclax schedules.
CR/Cri rate of AZA based and LDAC based, in P53 subset | Through study completion: 2 years after the last patient has been enrolled into the study, an average of 48 months.
  CR/CRi rate of AZA based and LDAC based triple combination with Quizartinib and Venetoclax schedules.
CR/Cri rate of AZA based and LDAC based, in IDH1/IDH2 subset | Through study completion: 2 years after the last patient has been enrolled into the study, an average of 48 months.
  CR/CRi rate of AZA based and LDAC based triple combination with Quizartinib and Venetoclax schedules.
MRD negativity rate in the BM | After cycle 1, cycle 4 and then every 3 cycles, being each cycle of 28 days.
  To evaluate the MRD negativity rate in the BM using MPFC and NGS-MRD, as part of analysis of biomarkers.
MRD negativity rate in PB | After cycle 1, cycle 4 and then every 3 cycles, being each cycle of 28 days.
  To evaluate the MRD negativity rate in PB using NGS-MRD, as part of analysis of biomarkers.
Natural Killer (NK) cell phenotypes and functions (immune recovery) analysis. | At screening and after first and fourth cycles of treatment, being each cycle of 28 days.
  Natural Killer (NK) substudy to analyse NK cell phenotypes and functions, as part of biomarker analysis.
Baseline and relapse molecular characterization by NGS. | At baseline and at through study completion due to relapse/resistance, an average of 48 months.
  Baseline and relapse molecular characterization by next generation sequencing (NGS), as part of biomarker analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Pau Montesinos, MD, Principal Investigator — Hospital Universitario La Fe; Juan Bergua, MD, Principal Investigator — Hospital San Pedro Alcántara; Carmen López-Carrero García, Study Chair — Fundación PETHEMA
Locations (15):
- Spain (15):
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares
  - Hospital Clínic, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario de Jerez de La Frontera, Jerez de la Frontera
  - Hospital de León (Complejo Asistencial Universitario de León), León
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Zarzuela, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital de Sant Joan de Deu (Manresa), Manresa
  - Hospital Clinico Universitario Virgen de La Arrixaca, Murcia
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitari Mutua de Terrassa, Terrassa
  - Hospital Universitario y Politécnico La Fe, Valencia

REFERENCES:
- [Background] Dohner H, Estey E, Grimwade D, Amadori S, Appelbaum FR, Buchner T, Dombret H, Ebert BL, Fenaux P, Larson RA, Levine RL, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz M, Sierra J, Tallman MS, Tien HF, Wei AH, Lowenberg B, Bloomfield CD. Diagnosis and management of AML in adults: 2017 ELN recommendations from an international expert panel. Blood. 2017 Jan 26;129(4):424-447. doi: 10.1182/blood-2016-08-733196. Epub 2016 Nov 28. PMID 27895058
- [Background] Juliusson G, Antunovic P, Derolf A, Lehmann S, Mollgard L, Stockelberg D, Tidefelt U, Wahlin A, Hoglund M. Age and acute myeloid leukemia: real world data on decision to treat and outcomes from the Swedish Acute Leukemia Registry. Blood. 2009 Apr 30;113(18):4179-87. doi: 10.1182/blood-2008-07-172007. Epub 2008 Nov 13. PMID 19008455
- [Background] Menzin J, Lang K, Earle CC, Kerney D, Mallick R. The outcomes and costs of acute myeloid leukemia among the elderly. Arch Intern Med. 2002 Jul 22;162(14):1597-603. doi: 10.1001/archinte.162.14.1597. PMID 12123403
- [Background] Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Santini V, Gattermann N, Germing U, Sanz G, List AF, Gore S, Seymour JF, Dombret H, Backstrom J, Zimmerman L, McKenzie D, Beach CL, Silverman LR. Azacitidine prolongs overall survival compared with conventional care regimens in elderly patients with low bone marrow blast count acute myeloid leukemia. J Clin Oncol. 2010 Feb 1;28(4):562-9. doi: 10.1200/JCO.2009.23.8329. Epub 2009 Dec 21. PMID 20026804
- [Background] Burnett AK, Milligan D, Prentice AG, Goldstone AH, McMullin MF, Hills RK, Wheatley K. A comparison of low-dose cytarabine and hydroxyurea with or without all-trans retinoic acid for acute myeloid leukemia and high-risk myelodysplastic syndrome in patients not considered fit for intensive treatment. Cancer. 2007 Mar 15;109(6):1114-24. doi: 10.1002/cncr.22496. PMID 17315155
- [Background] Cortes JE, Kantarjian H, Foran JM, Ghirdaladze D, Zodelava M, Borthakur G, Gammon G, Trone D, Armstrong RC, James J, Levis M. Phase I study of quizartinib administered daily to patients with relapsed or refractory acute myeloid leukemia irrespective of FMS-like tyrosine kinase 3-internal tandem duplication status. J Clin Oncol. 2013 Oct 10;31(29):3681-7. doi: 10.1200/JCO.2013.48.8783. Epub 2013 Sep 3. PMID 24002496
- [Background] Martinelli G, Perl AE, Dombret H, et al. Effect of quizartinib (AC220) on response rates and long-term survival in elderly patients with FLT3-ITD positive or negative relapsed/refractory acute myeloid leukemia. J Clin Oncol. 2013;31 (suppl): abstr 7021
- [Background] Konopleva M, Contractor R, Tsao T, Samudio I, Ruvolo PP, Kitada S, Deng X, Zhai D, Shi YX, Sneed T, Verhaegen M, Soengas M, Ruvolo VR, McQueen T, Schober WD, Watt JC, Jiffar T, Ling X, Marini FC, Harris D, Dietrich M, Estrov Z, McCubrey J, May WS, Reed JC, Andreeff M. Mechanisms of apoptosis sensitivity and resistance to the BH3 mimetic ABT-737 in acute myeloid leukemia. Cancer Cell. 2006 Nov;10(5):375-88. doi: 10.1016/j.ccr.2006.10.006. PMID 17097560
- [Background] Tsao T, Shi Y, Kornblau S, Lu H, Konoplev S, Antony A, Ruvolo V, Qiu YH, Zhang N, Coombes KR, Andreeff M, Kojima K, Konopleva M. Concomitant inhibition of DNA methyltransferase and BCL-2 protein function synergistically induce mitochondrial apoptosis in acute myelogenous leukemia cells. Ann Hematol. 2012 Dec;91(12):1861-70. doi: 10.1007/s00277-012-1537-8. Epub 2012 Aug 15. PMID 22893484
- [Background] Nakayama K, Nakayama K, Negishi I, Kuida K, Sawa H, Loh DY. Targeted disruption of Bcl-2 alpha beta in mice: occurrence of gray hair, polycystic kidney disease, and lymphocytopenia. Proc Natl Acad Sci U S A. 1994 Apr 26;91(9):3700-4. doi: 10.1073/pnas.91.9.3700. PMID 8170972
- [Background] Yamamura K, Kamada S, Ito S, Nakagawa K, Ichihashi M, Tsujimoto Y. Accelerated disappearance of melanocytes in bcl-2-deficient mice. Cancer Res. 1996 Aug 1;56(15):3546-50. PMID 8758925
- [Background] Lees JA, Weinberg RA. Tossing monkey wrenches into the clock: new ways of treating cancer. Proc Natl Acad Sci U S A. 1999 Apr 13;96(8):4221-3. doi: 10.1073/pnas.96.8.4221. No abstract available. PMID 10200241
- [Background] Shapiro GI. Cyclin-dependent kinase pathways as targets for cancer treatment. J Clin Oncol. 2006 Apr 10;24(11):1770-83. doi: 10.1200/JCO.2005.03.7689. PMID 16603719
- [Background] Schwartz GK, Shah MA. Targeting the cell cycle: a new approach to cancer therapy. J Clin Oncol. 2005 Dec 20;23(36):9408-21. doi: 10.1200/JCO.2005.01.5594. PMID 16361640
- [Background] Chen YN, Sharma SK, Ramsey TM, Jiang L, Martin MS, Baker K, Adams PD, Bair KW, Kaelin WG Jr. Selective killing of transformed cells by cyclin/cyclin-dependent kinase 2 antagonists. Proc Natl Acad Sci U S A. 1999 Apr 13;96(8):4325-9. doi: 10.1073/pnas.96.8.4325. PMID 10200261
- [Background] Cheson BD, Bennett JM, Kopecky KJ, Buchner T, Willman CL, Estey EH, Schiffer CA, Doehner H, Tallman MS, Lister TA, Lo-Coco F, Willemze R, Biondi A, Hiddemann W, Larson RA, Lowenberg B, Sanz MA, Head DR, Ohno R, Bloomfield CD; International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. Revised recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. J Clin Oncol. 2003 Dec 15;21(24):4642-9. doi: 10.1200/JCO.2003.04.036. PMID 14673054
- [Background] Creutzig U, Kaspers GJ. Revised recommendations of the International Working Group for diagnosis, standardization of response criteria, treatment outcomes, and reporting standards for therapeutic trials in acute myeloid leukemia. J Clin Oncol. 2004 Aug 15;22(16):3432-3. doi: 10.1200/JCO.2004.99.116. No abstract available. PMID 15310791
- [Background] European Medicines Agency. Summary of product characteristics. https://www.ema.europa.eu/documents/product-information/vidaza-epar-product-information_en.pdf. Accessed 12 December 2018
- [Background] CIMA- Centro de información online de medicamentos de la AEMPS - https://cima.aemps.es/cima/pdfs/es/ft/49154/FT_49154.pdf
- [Background] U.S. Department of Health and Human Services. National Institutes of Health. National Cancer Institute. https://evs.nci.nih.gov/ftp1/CTCAE/CTCAE_4.03/CTCAE_4.03_2010-06-14_QuickReference_5x7.pdf. Accessed 12 December 2018
- [Background] Montesinos P, Lorenzo I, Martin G, Sanz J, Perez-Sirvent ML, Martinez D, Orti G, Algarra L, Martinez J, Moscardo F, de la Rubia J, Jarque I, Sanz G, Sanz MA. Tumor lysis syndrome in patients with acute myeloid leukemia: identification of risk factors and development of a predictive model. Haematologica. 2008 Jan;93(1):67-74. doi: 10.3324/haematol.11575. PMID 18166787
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] European Organization for Research and Treatment of Cancer QLQ-C30 questionnaire (EORTC Quality of Life): https://www.eortc.org/app/uploads/sites/2/2018/08/Specimen-QLQ-C30-English.pdf.